CLINICAL TRIAL: NCT01373060
Title: A Double-blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Oral Doses of ASP1941 in Healthy Male Taiwanese Subjects
Brief Title: A Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of ASP1941 in Healthy Male Taiwanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 1941-CL-2001
Record Dates: First submitted 2011-05-31; First posted 2011-06-14 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Healthy; Pharmacokinetics of ASP1941
Keywords: ASP1941; ipragliflozin; plasma glucose; urine glucose
MeSH Terms: conditions — Glycosuria | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP1941 group (Experimental)
  Interventions: Drug: ASP1941
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP1941 — oral
  Other Names: ipragliflozin
  Arms: ASP1941 group
Drug: Placebo — oral
  Arms: placebo group

SUMMARY:
This study assesses the safety, tolerability, pharmacokinetics and pharmacodynamics of ASP1941 orally administered as single doses to healthy adult male Taiwanese subjects.

DETAILED DESCRIPTION:
The subjects will be administered a single dose of ASP1941 or placebo under fasting condition. Plasma and urine levels of ASP1941 and glucose will be measured to investigate pharmacokinetic and pharmacodynamic properties of ASP1941.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 50 and 85 kg, and Body Mass Index (BMI) between 17.6 and 26.4 kg/m2 inclusive

Exclusion Criteria:

* Medical history of metabolic disease, hepatic disease, heart disorder, respiratory disease, gastrointestinal disease, renal disease, cerebrovascular disorder, malignant tumor, drug allergy and drug/alcohol dependence
* Blood pressure, pulse rate, body temperature and 12-lead ECG are outside of the preset normal range
* Labo test results deviate from preset normal range
* Receiving treatment, including medication, within 14 days before the study
* Receiving medication in another clinical study or a post-marketing clinical trial within 3 months before the study
* Donates 500mL of whole blood within 3 months or 250mL within 2 months or blood components within 14 days before the study
* Drinking more than 45g of alcohol, or smoking more than 20 cigarettes per day
* Employed by the sponsor, delegated CRO or the study site
* Fasting plasma glucose level of < 70 mg/dL or ≥110 mg/dL or with an HbA1c ≥5.8%
* Subjects with positive serology test for Hepatitis B antigen, Hepatitis A virus IgM, anti-Hepatitis C virus or anti-Human Immunodeficiency virus-1 or -2

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety assessed by the incidence of adverse events, vital signs, safety lab tests and 12-lead ECG | up to 72 hours

SECONDARY OUTCOMES:
Cmax of ASP1941 plasma concentration | up to 72 hours
AUC (Area under the curve) of ASP1941 plasma concentration | up to 72 hours
Changes in plasma glucose | baseline and up to 72 hours
Changes in urine glucose | baseline and up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Taipei, Taiwan